CLINICAL TRIAL: NCT00977600
Title: A Randomized, Crossover, Open-label Phase 1 Study of Glyceryl Tri-(4-phenylbutyrate) (GT4P)
Brief Title: A Study of Glyceryl Tri-(4-phenylbutyrate) (GT4P)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Ucyclyd Pharma, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UP 1204-001
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Ammonul; Sodium phenylacetate; sodium benzoate; Buphenyl; sodium phenylbutyrate; HPN-100; GT4P; Glyceryl tri-(4-phenylbutyrate); Healthy Volunteers
MeSH Terms: interventions — glycerol phenylbutyrate; ammonul; 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GT4P-F (Experimental): GT4P-F (80% GT4P) was supplied as an odorless, colorless, tasteless liquid oil in 125 ml bottles. This formulation was designed to be mixed in water and create a self-emulsifying suspension, thus administered in water for the trial. The administered dose was calculated to contain the number of moles of PBA equivalent to 3 g/m2 of PBA. GT4P-F was mixed in 50 ml of water, taken orally, and then the cup rinsed with 50 ml of water and taken orally. GT4P-F was stored at ambient temperature away from light.
  Interventions: Drug: HPN-100
- GT4P-API (Experimental): GT4P-API was supplied as an odorless, colorless, tasteless oil in 125 ml bottles. The administered dose was calculated to contain the number of moles of PBA equivalent to 3 g/m2 of PBA. GT4P-API was taken orally and washed down with 100 ml of water. GT4P-API was stored at ambient temperature, away from light.
  Interventions: Drug: HPN-100
- Ammonul (Active Comparator): Ammonul® was supplied as single-use glass vials of 10% sodium phenylacetate and 10% sodium benzoate for intravenous injection. Ammonul® was diluted before use with sterile dextrose injection 10% to a concentration of 9 mg/ml. Once diluted it was kept at room temperature and used within 24 hours. The dose was 2.75 g/m2 and was administered as an intravenous infusion over a 120-minute period. Ammonul® was stored at 25°C, within a range of 15-30°C.
  Interventions: Drug: Ammonul
- Buphenyl (Active Comparator): Sodium phenylbutyrate or Buphenyl® was supplied as a white powder in 250 g bottles. The required amount of powder (equivalent to 3 g/m2 of PBA) was weighed out, mixed in 100 ml of water, and administered orally. Doses were calculated on a weight/volume basis and corrected for sodium content and purity. Buphenyl® was stored at ambient temperature.
  Interventions: Drug: Buphenyl

INTERVENTIONS:
Drug: HPN-100 — HPN-100 is a triglyceride that has a similar mechanism of action as Buphenyl. It is a liquid with minimal taste and odor. HPN-100 is broken down to phenylbutyric acid (PBA). PBA is converted to phenyl acetic acid (PAA) that is the active metabolite. Three teaspoons of HPN-100 (~17.4mL) delivers equivalent amount of PBA that 40 tablets of NaPBA do.
  Arms: GT4P-API; GT4P-F
Drug: Ammonul
  Arms: Ammonul
Drug: Buphenyl
  Arms: Buphenyl

SUMMARY:
To determine the safety and tolerability of single oral doses of HPN-100 as a formulation (GT4P-F) and GT4P as the active pharmaceutical ingredient (GT4P-API) administered to healthy male subjects.

DETAILED DESCRIPTION:
A randomized, open-label, four-treatment, four-period crossover study in which healthy male subjects received a single dose of each of the following four treatments on four separate dosing days, 7 days apart:

* Oral sodium phenylbutyrate (Buphenyl®) equivalent to 3 g/m2 of 4-phenylbutyric acid (PBA) per dose
* Oral GT4P-F mole equivalents to 3 g/m2 of PBA per dose
* Oral GT4P-API mole equivalents to 3 g/m2 of PBA per dose
* Intravenous 10% sodium phenylacetate plus 10% sodium benzoate (Ammonul®) 2.75 g/m2

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

Subjects were required to fulfill the following criteria in order to participate in the study:

* Males aged 18 to 45 years of age
* Ability to provide written, informed consent before any study-related procedures, and ability, in the opinion of the investigator, to comply with all the requirements of the study
* Subjects who were in good health as determined by a medical history, physical examination, serum chemistry, hematology, urinalysis, 12 lead ECG, and vital signs
* Weight within the range of 60-120 kg

Exclusion Criteria:

Subjects who fulfilled any of the following criteria were excluded from the study:

* Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurologic, immunologic, or psychiatric disorder(s), as determined by the investigator
* Clinically significant abnormal laboratory values (as determined by the investigator)
* Significant illness within 14 days prior to screening
* Any disorder that might significantly interfere with the absorption, distribution, metabolism, or excretion of any drug
* Use of any prescription medication within 14 days prior to screening
* Use of dietary supplements, herbal medicines, vitamins, or over-the-counter medication(s) (with the exception of acetaminophen ≤ 500 mg/day) within 10 days prior to first dosing
* Positive drugs of abuse urine test at screening or pre-dose day (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, methadone)
* Positive alcohol breath test at screening or pre-dose day
* Donation or loss of blood (500 ml or more) within 30 days prior to first dosing, or during the study
* Donation or loss of plasma within 7 days prior to first dosing, or during the study
* History of or current hepatitis or carriers of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies (anti-HC)
* History of acquired immunodeficiency syndrome (AIDS) or determined HIV positive at screening
* Use of any investigational drug within 12 weeks prior to first dosing
* Known hypersensitivity to sodium phenylbutyrate or similar drugs
* Previous exposure to sodium phenylbutyrate

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The rate of adverse events | 33 Days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Medical Sanitary Division #2, Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] McGuire BM, Zupanets IA, Lowe ME, Xiao X, Syplyviy VA, Monteleone J, Gargosky S, Dickinson K, Martinez A, Mokhtarani M, Scharschmidt BF. Pharmacology and safety of glycerol phenylbutyrate in healthy adults and adults with cirrhosis. Hepatology. 2010 Jun;51(6):2077-85. doi: 10.1002/hep.23589. PMID 20512995